CLINICAL TRIAL: NCT01910142
Title: The Effect of Nutritional Intervention on Bone Metabolism as Assessed by 41Ca and Modeling; Proof of Concept
Brief Title: Effect of Nutrition on Bone Metabolism as Assessed by 41Ca
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Principal Investigator, Henk FJ Hendriks, PhD, TNO
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 8145
Record Dates: First submitted 2010-04-09; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Osteoporosis
Keywords: bone metabolism
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin K; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- calcium supplement with vitamin K (Active Comparator): Milk product supplying about 420 mg Ca and 7.5 μg vitamin D3 and 100 μg vitamin K. Additional 200 mg calcium in the form of carbonate
  Interventions: Dietary Supplement: vitamin K; Dietary Supplement: calcium
- calcium supplement without vitamin K (Placebo Comparator): Milk product supplying about 420 mg Ca and 7.5 μg vitamin D3. no vitamin K. Additional 200 mg calcium in the form of carbonate
  Interventions: Dietary Supplement: calcium

INTERVENTIONS:
Dietary Supplement: vitamin K — A calcium product will be given either with or without vitamin K. Each intervention will last for 5 weeks, each followed by a 5 week wash-out. The first intervention will start about 4 months after inclusion and the single 41Ca bolus.
  Arms: calcium supplement with vitamin K
Dietary Supplement: calcium

SUMMARY:
The present study aims to develop a technique based on a single dose of a calcium isotope, which enables to determine the effect of a nutritional intervention on bone calcium metabolism. For this purpose nutritional interventions with calcium, vitamin D and vitamin K will be applied in postmenopausal women. Treatment effects will be determined by the urinary excretion of the calcium isotope and related to classical bone markers.

DETAILED DESCRIPTION:
In the present proposal a method is described that may enable studying the effect of nutrition on bone calcium turnover far more accurate, within a shorter time frame and therefore less intensive for the volunteers in clinical studies as compared to presently existing methods. This method will enable screening for promising food concepts for combating osteoporosis within a relatively short time. Recent developments show that use of the nuclide 41Calcium (41Ca) and measurement by accelerator mass spectrometry (AMS) has great potential in measuring effects on bone level within a relatively short period of time. When introducing a diet change (intervention) the bone metabolism of calcium may change resulting in a changed 41Ca-signal in the urine. So far a few medication studies with osteoporotic volunteers have been performed and it appears that this ultrahigh sensitive technique may also be applicable for nutrition studies in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire,
   * physical examination
   * results of the pre-study laboratory tests
2. Females aged 50-68 years at Day 01 of the study
3. Relatively low calcium intake as assessed by dairy intake questionnaire
4. Body Mass Index (BMI) < 30 kg/m2
5. Postmenopausal as confirmed by Follicle stimulating hormone (FSH) and oestradiol (E2) blood levels (FSH > 40IU/L, E2 < 70 pg/mL)
6. Normal Dutch eating habits
7. Voluntary participation
8. Having given written informed consent
9. Willing to comply with the study procedures
10. Appropriate veins for blood sampling/cannula insertion according to TNO
11. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
12. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease or hypertension and gastrointestinal disease
4. Prescribed medication, including hormone replacement therapy (within 6 months before start of the study) and anticoagulant medication.
5. Reported intolerance for dairy products
6. Not willing to stop the use of Boerenkarnemelk and cheese of the following Dutch brands: Emmenthaler, Gruyere, Leer/Maasdammer
7. Alcohol consumption > 21 units/week
8. Not willing to stop use of supplements containing minerals or vitamins
9. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
10. Reported slimming or medically prescribed diet
11. Reported vegan, vegetarian or macrobiotic
12. Recent blood donation (<1 month prior to the start of the study)
13. Not willing to give up blood donation during the study.
14. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
15. Not having a general practitioner
16. Not willing to accept information-transfer concerning participation in the study, or information regarding her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from her general practitioner.

Ages: 50 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
urinary 41calcium excretion | on study day numbers: 36, 71, 106, 113, 120, 127, 134, 141, 148, 155, 162, 169, 176, 183, 190, 197, 204, 211, 218, 225, 232, 239, 246, 253, 260, 267, 274, 281, 288
  Urine is collected for measurement of 41Ca. The concentration change of 41Ca during the intervention period indicates the efficacy of the intervention.

SECONDARY OUTCOMES:
commonly accepted biomarkers for bone metabolism | on study day numbers: 148, 183, 218, 253, 288
  Plasma osteocalcin and urinary deoxypyridinolin/creatinin ratio are measured as traditional markers for bone accretion and bone resorption respectively. These are the most commonly used biomarkers for bone metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Gertruud C Bakker, PhD, Principal Investigator — TNO